CLINICAL TRIAL: NCT03810131
Title: Study Protocol for a Feasibility Study of a Novel ACT-based eHealth Psychoeducational Intervention for Students With Mental Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, Darren Edwards, Principle Investigator, Swansea University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEdwards
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: A Bite of ACT' (BOA) Acceptance and Commitment Therapy Online Psychoeducation Course; A Wait-list Control
Keywords: Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control (No Intervention): This is a group who are waiting for treatment (the control group)
- BOA online intervention (Experimental): The is the group who are receiving the BOA online intervention.
  Interventions: Other: 'A Bite of ACT' (BOA)

INTERVENTIONS:
Other: 'A Bite of ACT' (BOA) — An online Acceptance and Commitment Therapy transdiagnostic psychoeducational intervention called 'A Bite of ACT' (BOA)
  Arms: BOA online intervention

SUMMARY:
Here we propose a protocol for assessing the feasibility and acceptability of a randomised controlled trial (RCT) of an online transdiagnostic psychoeducational intervention called 'A Bite of ACT' (BOA) compared to a waitlist control.

DETAILED DESCRIPTION:
Introduction: Recent studies reveal a high prevalence of depression, anxiety, and stress symptoms among university students, highlighting an urgent need for preventative measures at low cost to better support often overwhelmed support services.

Objectives: Here we propose a protocol for assessing the feasibility and acceptability of a randomised controlled trial (RCT) of an online transdiagnostic psychoeducational intervention called 'A Bite of ACT' (BOA) compared to a waitlist control.

Methods and analysis:

A randomised controlled trial with crossover design will be conducted at baseline, and two follow-up periods. The primary outcome measure will be the ACCEPT checklist, while secondary outcomes include measures of wellbeing, depression, anxiety, and stress (DASS21) and a process measure (psychological flexibility AAQII). Qualitative interviews and preliminary health economics analysis will provide additional insights. Analysis will focus on descriptive statistics and feasibility outcomes and calculate a treatment effect size to determine sample size needed for any future trial (if indicated).

ELIGIBILITY:
Inclusion Criteria:

- 1. Participants will be included in the study if they report any feelings of depression, anxiety, and stress (regardless of severity). Participants with an existing psychological disorder will be eligible for the study as long as they are receiving treatment for the disorder and that this treatment does not change over the duration of the study proposed here. Clear instructions will be provided indicating that our BOA intervention should not be used as an alternative to GP/NHS prescribed medication or psychological interventions such as CBT.

2. Participants will need normal or corrected to normal vision and to be able to read and write English.

Exclusion Criteria:

- 1. Participants will be excluded if they do not have mental distress as stated above.

2. Participants will be excluded if they do not have normal or corrected to normal vision and to be able to read and write English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Acceptance Checklist for Clinical Effectiveness Pilot Trials (ACCEPT) (Charlesworth, Burnell, Hoe, Orrell, & Russell, 2013) | One years (anticipated)
  Acceptance Checklist for Clinical Effectiveness Pilot Trials (ACCEPT)

SECONDARY OUTCOMES:
Depression Anxiety Stress Scales | One years (anticipated)
  Depression Anxiety Stress Scales (short-form DASS-21). This is the short version of this measure and is a general psychological distress measure with good construct validity (confirmatory factor analysis of 0.94). It has good internal reliability as measured through Cronbach's alpha coefficients, which are 0.88 for depression, 0.82 for anxiety, 0.90 for stress and 0.93 for the total scale (Henry & Crawford, 2005).
Social connectedness | One years (anticipated)
  Social connectedness (adapted from Russell's (1996) UCLA Loneliness Scale (Kok et al., 2013). This includes two questions; (1) "During these social interactions, I felt 'in tune' with the person/s around me", and (2) "During these social interactions, I felt close to the person/s." Responses are made on a 7-point scale (1 = not at all true, 7 = very true). The Cronbach's alpha coefficients for these two items ranged from .80 to .98 (M = .94, SD = .03) (Kok et al., 2013).
EuroQol five dimensions | One years (anticipated)
  EuroQol five dimensions (EQ5D). The EQ5D is a measure for health-related quality of life (HRQOL) statues. Within it, there are five components which assess mobility, self-care, usual activities, pain and discomfort, as well as anxiety. It also has a visual analogue scale (VAS) for measuring current health status. Scores for these will be calculated for each of these five subsections as well as including the VIS and total EQ5D score of all five subsections. The EQD5 correlates well with other health related questionnaires such as the SF-36 (r = 0.61, p<0.0001) and PDQ-39 (r = -0.75, p<0.0001) (Schrag, Selai, Jahanshahi, & Quinn, 2000).
Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) | One years (anticipated)
  Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) (Tennant et al., 2007). Is a measure of mental well-being with a focus on positive aspects of mental health. It has good internal consistency with a Cronbach's alpha coefficient of 0.89 (student sample) and 0.91 (general population sample).

OTHER OUTCOMES:
Heart rate variability (HRV) | One years (anticipated)
  Heart rate variability (HRV). This measures the beat-to-beat variation of the R-R intervals of the electrocardiogram recording and is controlled via the sympathetic and parasympathetic components of the autonomic nervous system (ANS). This is a commonly indexed measure of vagal function and important mediator of health and wellbeing associated with emotion regulation and longevity (Kemp, Arias, et al., 2017) . Measurement of the HRV to assess autonomic changes can be performed using a sensitive and non-invasive technique through an electrocardiogram.
Mindfulness Attention Awareness Scale (MAAS) | One years (anticipated)
  Mindfulness Attention Awareness Scale (MAAS). This is a 15-item scale and is used to measure participant's awareness of moment to moment experiences. This mindful self-awareness can be improved through practicing mindfulness. Also, the absence of this skill correlates with decreased self-awareness (Brown & Ryan, 2003). The scale is rated from 1 (almost always) to 6 (almost never) and are then averaged. The internal validity of the MAAS is high where a Cronbach's alpha coefficient of 0.83 has been reported (Frewen, Evans, Maraj, Dozois, & Partridge, 2008).
Acceptance and Action Questionnaire | One years (anticipated)
  Acceptance and Action Questionnaire- second version (AAQ-II). This is a 10 item scale, developed by (Bond et al., 2011) to measure psychological flexibility which involves the ability to accept and be open to difficult thoughts and feelings as well as engage in valued behaviour in the presence of the difficult thoughts and feelings. Higher scores indicate higher psychological flexibility, and the measure has good construct validity with a Cronbach's alpha coefficient of 0.84 (Bond et al., 2011).

CONTACTS AND LOCATIONS:
Locations (1):
- Swansea University, Swansea, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edwards DJ, Rainey E, Boukouvala V, Wells Y, Bennett P, Tree J, Kemp AH. Novel ACT-based eHealth psychoeducational intervention for students with mental distress: a study protocol for a mixed-methodology pilot trial. BMJ Open. 2019 Jul 16;9(7):e029411. doi: 10.1136/bmjopen-2019-029411. PMID 31315873